CLINICAL TRIAL: NCT05141552
Title: The Safety of Dapagliflozin in Hemodialysis Patients With Heart Failure
Acronym: SDHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Leyi Gu, Professor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KY2021-162
Record Dates: First submitted 2021-11-07; First posted 2021-12-02 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Hemodialysis Complication
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dapa group (Experimental): subjects will be treated with dapagliflozin (10mg per day) and standard anti-heart failure therapy (including RAS inhibitors, beta-blocker, Aldosterone inhibitors)
  Interventions: Drug: Dapagliflozin 10Mg Tab
- control group (No Intervention): subjects will be treated with standard anti-heart failure therapy (including RAS inhibitors, beta-blocker, Aldosterone inhibitors)

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — In both group, subjects keep blood purification and anti heart failure treatment, including ARNI, RASi, Aldosterone inhibitors and beta receptor blocker.
  Other Names: Control
  Arms: dapa group

SUMMARY:
SGLT2 inhibitor is a new type of sugar-lowering medicine and is recommended to treat heart failure. eGFR lower than 30ml/min/1.73M2 is contraindication of SGLT2 inhibitor. Heart failure is one of the most frequency CVD events for hemodialysis patients. But hemodialysis patient is unable to be treated with SGLT2 inhibitors as the contraindication. However, solute and fluid clearance are dependent on dialysis, but not renal function in hemodialysis patients. There is no data of SGLT2 inhibitor on hemodialysis patients. The aim of the present study is evaluate the safety of Dapagliflozin in hemodialysis patients with heart failure.

This is a randomized, control, open study. 20 hemodialysis patients with heart failure will be recruited. 10 of 20 subjects will be treated with dapagliflozin 10mg everyday for 12 weeks. The primary outcome is the number of patients with hypoglycemia or urinary infection. The secondary outcomes is the changes of NT-.

DETAILED DESCRIPTION:
Evaluate the safety of dapagliflozin in hemodialysis patients with heart failure is the main purpose of this study. and Estimate the change of NT-proBNP is the secondary purpose.

This is a randomized, control and open study.

The including criteria are 1. Understand the present study and sign informed consert 2. Age is between 18 and 70 3. 2 or 3 times blood purification treatments (inclusion hemodialysis, hemofiltration, hemoperfusion) every week, 4. Blood purification treatment more than 3 month 5. Using AV fistula or artificial vascular access 6. With chronic heart failure (NYHC II-IV), and NT-proBNP>11500 or BNP>500 7. ARNI or RAS inhibitor or Aldosterone inhibitors treatment for at least 4 weeks with a stable dose The exclusion criteria are 1.Blood purification less than 3 month 2.With fluid overload and URR<50% 3.Have severe hypoglycemia (more than 2 events with 4 weeks prior to sign concert information) 4.Have severe hypotension (blood pressure <90/60mmHg more than 3 times with 4 weeks prior to sign concert information) 5.Have acute pulmonary edema 6.Have ketoacidosis 7.Have active pyelnephritis and symptomatic lower urinary infection 8.Subject is pregnant , is breast feeding 9.Subject has known SGLT2 inhibitor allergy or intolerance adverse reactions 10.Subject is currentluy enrolled in or has not yet completed at least 30days since ending other investigational device or drug trials 11.Investigator believe subject is not suitable for this study

Subjects will divide into two groups. Dapa group will be treated with dapagliflozin 10mg qd and standard anti-heart failure therapy. Control group will be treated with standard anti-heart failure therapy.

The primary outcome is the number of patients with hypoglycemia or urinary tract infection. The secondary outcome is the change of NT-proBNP

ELIGIBILITY:
Inclusion Criteria:

1. Understand the present studyAgree and sign informed consert
2. Age is between 18 and 70 Men or women ≧18 years and <70 years of age at screening
3. Treated with maintenance blood purification 2 or 3 times blood purification treatments (including hemodialysis, hemofiltration, hemoperfusion) every week2 or 3 times a week,
4. Blood purification treatment more than 3 month before randomization
5. Blood purification by uUsing AV fistula or artificial vascular access
6. DiagnosisWith chronic heart failure (NYHC II-IV), and NT-proBNP>11500 or BNP>500
7. ARNI or RAS inhibitor or Aldosterone inhibitors or beta receptor blocker treatment for at least 4 weeks with a stable dose.

Exclusion Criteria:

1. Blood purification less than 3 month
2. With fluid overload and URR<50%
3. Have severe hypoglycemia (more than 2 events with 4 weeks prior to sign concert information)
4. Have severe hypotension (blood pressure <90/60mmHg more than 3 times with 4 weeks prior to sign concert information)
5. Have acute pulmonary edema
6. Have ketoacidosis
7. Have active pyelnephritis and symptomatic lower urinary infection
8. Subject is pregnant , is breast feeding
9. Subject has known SGLT2 inhibitor allergy or intolerance adverse reactions
10. Subject is currentluy enrolled in or has not yet completed at least 30days since ending other investigational device or drug trials
11. Investigator believe subject is not suitable for this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
the number of patients with hypoglycemia or urinary tract infection | 12 weeks
  the number of patients with hypoglycemia or urinary tract infection

SECONDARY OUTCOMES:
Change of NT-proBNP | 12 weeks
  Change of NT-proBNP

CONTACTS AND LOCATIONS:
Overall Officials: Leyi Gu, Principal Investigator — RenJi Hospital
Locations (1):
- Department of nephrology , Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Result] Packer M, Anker SD, Butler J, Filippatos G, Pocock SJ, Carson P, Januzzi J, Verma S, Tsutsui H, Brueckmann M, Jamal W, Kimura K, Schnee J, Zeller C, Cotton D, Bocchi E, Bohm M, Choi DJ, Chopra V, Chuquiure E, Giannetti N, Janssens S, Zhang J, Gonzalez Juanatey JR, Kaul S, Brunner-La Rocca HP, Merkely B, Nicholls SJ, Perrone S, Pina I, Ponikowski P, Sattar N, Senni M, Seronde MF, Spinar J, Squire I, Taddei S, Wanner C, Zannad F; EMPEROR-Reduced Trial Investigators. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. N Engl J Med. 2020 Oct 8;383(15):1413-1424. doi: 10.1056/NEJMoa2022190. Epub 2020 Aug 28. PMID 32865377
- [Result] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Result] Singh M, Kumar A. Risks Associated with SGLT2 Inhibitors: An Overview. Curr Drug Saf. 2018;13(2):84-91. doi: 10.2174/1574886313666180226103408. PMID 29485006